CLINICAL TRIAL: NCT01146873
Title: Treatment Options for Protease Inhibitor-exposed Children
Acronym: NEVEREST-III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Witwatersrand, South Africa (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Louise Kuhn, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAE1145; R01HD061255 (NIH)
Record Dates: First submitted 2010-06-08; First posted 2010-06-22 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: HIV/AIDS; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — efavirenz; Lopinavir; Stavudine; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: Lopinavir/ritonavir (LPV/r) (Active Comparator): Participants are assigned to remain on their current LPV/r-based antiretroviral regimen. Ritonavir-boosted lopinavir syrup was given twice per day at 230 mg/m^2 per dose. Children able to swallow tablets were given 1 tablet twice per day (200 mg lopinavir/50 mg ritonavir) if body surface area was less than 0.9m^2 or 2 tablets twice per day if body surface area was 0.9m^2 or higher.
  Interventions: Drug: Lopinavir/ritonavir (LPV/r)
- Group 2: Efavirenz (EFV) (Experimental): Participants are assigned to switch to an EFV-based antiretroviral regimen. Efavirenz was prescribed once daily in the evening at 200 mg for weights of 10 kg to 13.9 kg (22-30 lb) and 300mg for weights of 14 kg to 24.9 kg (31-55 lb). Efavirenz was available in 50-mg and 200-mg capsules. If children were unable to swallow capsules, caregivers were shown how to open the capsules and dissolve the contents in water.
  Interventions: Drug: Efavirenz (EFV)
- Group D: Stavudine (D4T) (Active Comparator): Children are assigned to remain on their current antiretroviral regimen, which includes D4T. D4T was given at 1 mg/kg twice daily
  Interventions: Drug: Stavudine (D4T)
- Group A: Abacavir (ABC) (Experimental): Children stop taking D4T and switch to ABC. ABC was given at 8 mg/kg twice daily.
  Interventions: Drug: Abacavir (ABC)

INTERVENTIONS:
Drug: Efavirenz (EFV) — Children are assigned to begin a EFV-based antiretroviral based regimen.
  Arms: Group 2: Efavirenz (EFV)
Drug: Lopinavir/ritonavir (LPV/r) — Children are assigned to stay on their current LPV/r-based antiretroviral regimen.
  Arms: Group 1: Lopinavir/ritonavir (LPV/r)
Drug: Stavudine (D4T) — Children are assigned to stay on their current antiretroviral regimen which includes D4T.
  Arms: Group D: Stavudine (D4T)
Drug: Abacavir (ABC) — Children stop taking D4T and switch to ABC.
  Arms: Group A: Abacavir (ABC)

SUMMARY:
The investigators hypothesize that switching to a regimen based on efavirenz will be as effective and safe as remaining on a regimen based on Lopinavir/ritonavir for HIV-infected children.

The investigators propose an unblinded randomized clinical trial to evaluate a simplification, protease-inhibitor (PI)-sparing treatment strategy among nevirapine (NVP)-exposed HIV-infected children treated initially with lopinavir/ritonavir (LPV/r). HIV-infected children aged 3-5 years, who have a history of exposure to NVP as part of prevention of mother-to-child HIV transmission (PMTCT), initiated LPV/r-based therapy in the first 36 months of life or who were enrolled on the control arm of Neverest 2 and who are virally suppressed with a viral load < 50 copies/ml will be included. These children will be randomized to either substitute efavirenz (EFV) for LPV/r or to continue on their LPV/r-based regimen. Eight weeks prior to the primary randomization, eligible children will also be randomized to either remain on stavudine (D4T) or switch to abacavir (ABC). Children will be followed with regular viral load and other clinical tests for 48 weeks after the primary randomization. Children in the experimental arm who have breakthrough viremia (-defined as two subsequent viral loads > 1000 copies/ml) on the EFV-based regimen will reinitiate the LPV/r regimen. The primary objective is to test whether the durability of viral suppression is equivalent when children are switched to EFV-based therapy. The primary study endpoint is failure to have HIV RNA < 50 copies/ml and/or confirmed viremia >1000 copies/ml. Secondary aims include comparison of immune preservation, toxicities, selection of resistance mutations, and adherence across the two arms. Antiretroviral drug concentrations and adherence will be investigated as possible explanations for the success and/or failure of this simplification regimen. The overall goal of the study is to contribute to the evidence base to allow expansion of treatment options for HIV-infected children in low resource settings.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected child 3 to 5 years of age at time of screening for this trial if enrolled from outside or any age if enrolled from control arm of Neverest II.
* Reliable history or documented exposure to NVP used as part of PMTCT
* Initiated antiretroviral therapy with LPV/r at age less than 36 months
* Receiving LPV/r-based ART for at least 12 months
* At least one viral load measurement less than 50 copies/ml conducted as part of screening for the study
* ALT measurement grade I or less (DAIDS Toxicity Tables 2004) (Appendix A). These may be repeated until ALTs normalize if necessary.

Exclusion criteria:

* Prior treatment with any NNRTI drug as part of a therapeutic regimen
* Substitution of other NRTI drugs (instead of 3TC and D4T which are the standard first line regimen) will be allowed.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise Kuhn, PhD, Principal Investigator — Columbia University
Locations (1):
- Rahima Moosa Mother and Child Hospital, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Result] Coovadia A, Abrams EJ, Strehlau R, Shiau S, Pinillos F, Martens L, Patel F, Hunt G, Tsai WY, Kuhn L. Efavirenz-Based Antiretroviral Therapy Among Nevirapine-Exposed HIV-Infected Children in South Africa: A Randomized Clinical Trial. JAMA. 2015 Nov 3;314(17):1808-17. doi: 10.1001/jama.2015.13631. PMID 26529159
- [Derived] Murnane PM, Strehlau R, Shiau S, Patel F, Mbete N, Hunt G, Abrams EJ, Coovadia A, Kuhn L. Switching to Efavirenz Versus Remaining on Ritonavir-boosted Lopinavir in Human Immunodeficiency Virus-infected Children Exposed to Nevirapine: Long-term Outcomes of a Randomized Trial. Clin Infect Dis. 2017 Aug 1;65(3):477-485. doi: 10.1093/cid/cix335. PMID 28419200

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 300 study participants were recruited between June 2010 and October 2012.
Pre-assignment Details: Two children discontinued the study prior to randomization.
Period: Overall Study
Arm/Group | Group 1: Lopinavir/Ritonavir (LPV/r) | Group 2: Efavirenz (EFV)
Started | 148 | 150
Completed | 148 | 144
Not Completed | 0 | 6
Not completed — Transfer out | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Lopinavir/Ritonavir (LPV/r) | Group 2: Efavirenz (EFV) | Total
Number analyzed (Participants) | 148 | 150 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.26 (1.0) | 4.28 (0.9) | 4.27 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 78 | 158
  Male | 68 | 72 | 140

OUTCOME MEASURES:

1. Primary Outcome: Viral Rebound
Description: Probability of viral rebound defined as >=1 HIV RNA measurements >50 copies/ml using survival analysis by 48 weeks post-randomization.
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: probability of viral rebound
Groups:
- Group 1: Lopinavir/Ritonavir (LPV/r): Participants are assigned to remain on their current LPV/r-based antiretroviral regimen
- Group 2: Efavirenz (EFV): Participants are assigned to switch to an EFV-based antiretroviral regimen
Arm/Group | Group 1: Lopinavir/Ritonavir (LPV/r) | Group 2: Efavirenz (EFV)
Number analyzed (Participants) | 148 | 150
probability of viral rebound | 0.284 [0.211 to 0.357] | 0.176 [0.115 to 0.238]
Statistical Analysis 1: Comparison: Group 1: Lopinavir/Ritonavir (LPV/r) vs Group 2: Efavirenz (EFV); Test type: Non-Inferiority or Equivalence — The null hypothesis is that efavirenz is inferior to ritonavir-boosted lopinavir; p < 0.001, Kaplan-Meier methods; Risk Difference (RD) = 0.107

2. Primary Outcome: Viral Failure
Description: Probability of viral failure defined as >= 2 HIV RNA measurements >1000 copies/ml using survival analysis by 48 weeks post-randomization.
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: probability of viral failure
Arm/Group | Group 1: Lopinavir/Ritonavir (LPV/r) | Group 2: Efavirenz (EFV)
Number analyzed (Participants) | 148 | 150
probability of viral failure | 0.020 [0.002 to 0.043] | 0.027 [0.001 to 0.054]
Statistical Analysis 1: Comparison: Group 1: Lopinavir/Ritonavir (LPV/r) vs Group 2: Efavirenz (EFV); Test type: Non-Inferiority or Equivalence — The null hypothesis is that efavirenz is inferior to ritonavir-boosted lopinavir; p < 0.001, Kaplan-Meier methods; Risk Difference (RD) = -0.007

3. Secondary Outcome: CD4 Cell Percentage at 48 Weeks After Randomization
Description: CD4 Cell Percentage at 48 Weeks After Randomization
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | Group 1: Lopinavir/Ritonavir (LPV/r) | Group 2: Efavirenz (EFV)
Number analyzed (Participants) | 148 | 150
percentage of cells | 34.7 [33.6 to 35.8] | 37.5 [36.3 to 38.8]
Statistical Analysis 1: Comparison: Group 1: Lopinavir/Ritonavir (LPV/r) vs Group 2: Efavirenz (EFV); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Percentage of Participants With Elevated Total Cholesterol, Elevated LDL, Abnormal HDL, or Abnormal Triglycerides at 40 Weeks After Randomization
Description: Percentage of participants with elevated total cholesterol, elevated LDL, abnormal HDL, or abnormal triglycerides at 40 weeks after randomization
Time Frame: 40 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Lopinavir/Ritonavir (LPV/r) | Group 2: Efavirenz (EFV)
Number analyzed (Participants) | 148 | 150
percentage of participants
  Elevated total cholesterol | 24.8 | 13.3
  Elevated LDL | 18.6 | 9.8
  Abnormal HDL | 4.8 | 4.2
  Abnormal triglycerides | 22.8 | 10.5

5. Secondary Outcome: Highest Grade ALT After Randomization
Description: Highest grade ALT after randomization. Grading was determined based on the Division of AIDS (2004) Toxicity Tables to grade adverse reactions. Grading scale: 0 (none), 1 (mild), 2 (moderate), 3 (severe), 4 (potentially life-threatening).
Time Frame: through 48 weeks post randomization
Measure: Number; unit: number of participants
Arm/Group | Group 1: Lopinavir/Ritonavir (LPV/r) | Group 2: Efavirenz (EFV)
Number analyzed (Participants) | 148 | 150
number of participants
  Grade 0 | 139 | 120
  Grade 1 | 8 | 16
  Grade 2 | 0 | 10
  Grade 3 | 1 | 3
  Grade 4 | 0 | 1
Statistical Analysis 1: Comparison: Group 1: Lopinavir/Ritonavir (LPV/r) vs Group 2: Efavirenz (EFV); Test type: Superiority or Other; p = 0.003, Chi-squared

ADVERSE EVENTS:
Time Frame: Through 48 weeks after randomization
Arm/Group | Group 1: Lopinavir/Ritonavir (LPV/r) | Group 2: Efavirenz (EFV)
Serious Adverse Events (participants affected / at risk) | 0/148 | 2/150
Other Adverse Events (participants affected / at risk) | 0/148 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Lopinavir/Ritonavir (LPV/r) (N=148) | Group 2: Efavirenz (EFV) (N=150)
Seizure (Nervous system disorders) | 0 (0) | 2 — Seizures resolved after efavirenz was stopped and ritonavir-boosted lopinavir was restarted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other